CLINICAL TRIAL: NCT02347111
Title: A Prospective, Multi-Center, Randomized, Open Label Trial to Determine if a Common Atrial Fibrillation Risk Locus Modulates Differential Response to Antiarrhythmic Drugs
Brief Title: Pharmacogenetic Study of Antiarrhythmic Drugs for Atrial Fibrillation
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Dawood Darbar, MD, Professor of Medicine, University of Illinois at Chicago
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2018-1299
Record Dates: First submitted 2015-01-20; First posted 2015-01-27 (Estimated); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Flecainide; Sotalol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- flecainide 1st (Experimental): flecainide x 6 months, then crossover to sotalol x 6 months
  Interventions: Drug: Flecainide; Drug: Sotalol
- sotalol 1st (Experimental): sotalol x 6 months, then crossover to flecainide x 6 months
  Interventions: Drug: Flecainide; Drug: Sotalol

INTERVENTIONS:
Drug: Flecainide — flecainide up to 150mg twice daily for the control of atrial fibrillation
Drug: Sotalol — sotalol up to 120mg twice daily for the control of atrial fibrillation

SUMMARY:
In this pilot and feasibility study, the investigators will enroll patients with frequent symptomatic episodes of atrial fibrillation (AF) in a cross-over study testing two different classes of anti arrhythmic drugs (AADs). This pilot and feasibility study will provide preliminary data for a larger study in which the investigators will test the hypothesis that a common AF genetic risk allele modulates response to different AADs.

DETAILED DESCRIPTION:
1.0 Background

While atrial fibrillation (AF) is the most common sustained cardiac arrhythmia requiring therapy, it is also associated with increased risk of stroke, heart failure, myocardial infarction, dementia, and death. The number of Americans affected with AF is expected to surge to nearly 16 million by the year 2050. The AF epidemic may in part be related to the aging of the population and increasing prevalence of recently identified risk factors including obesity, metabolic syndrome, obstructive sleep apnea, and inflammation. Furthermore, there is increasing support for the idea that both common and rare genetic variants also increase susceptibility to AF which can clinically manifest in the presence of acquired risk factors. While clinical risk factors for AF are established, the genetic components of this "multiple-hit" genetic model for the development of AF have only recently been identified.

Despite recent advances in catheter-based and surgical therapies, anti-arrhythmic drugs (AADs) remain the mainstay of treatment for patients with symptomatic AF. However, response in an individual is highly variable with more than half of patients treated with AADs suffering a recurrence of AF within 6 to 12 months. The limited success of therapy for AF is related to poor understanding of the underlying pathophysiology, heterogeneity of the electrical and structural substrate, and the lack of targeted mechanism-based therapies. Thus, one major knowledge gap is predicting response to AADs in an individual patient. Contemporary membrane-active drugs used to suppress AF are incompletely and unpredictably effective and are associated with significant risks of proarrhythmia and non-cardiac toxicities. Furthermore, the current 'one-size fits all' approach to selecting AAD therapy for a patient with symptomatic AF is based largely on minimizing the risk of adverse events rather than on the likelihood of efficacy. Recent advances in our understanding of genetic mechanisms of AF support the overarching hypothesis we wish to test in future studies that variability in response to AAD therapy is modulated by common genetic variants associated with AF. Several AF susceptibility loci have been identified and validated in genome-wide association studies. In addition, we have shown that common AF risk single nucleotide polymorphisms (SNPs) at the chromosome (chr) 4q25 locus not only predict poor response to AADs but also recurrence of AF after ablation therapy and cardioversion.

While genetic approaches to AF have revealed that susceptibility to AF and response to therapy are modulated in part by the underlying genetic substrate, the translation of these discoveries to the bedside management of AF patients has thus far been limited. This relates to poor understanding of the underlying mechanisms associated with common AF risk alleles, challenges associated with determining efficacy of AADs and lack of genotype-directed prospective studies. Our preliminary data showed that a common chr4q25 SNP associated with AF predicted successful symptom control in patients treated with AADs and individuals who carried the risk variant responded better to Vaughan Williams class I vs. class III AADs. Based on the information collected in this feasibility and pilot study, we propose to conduct a prospective pharmacogenomic study where a cohort of patients with frequent symptomatic paroxysmal AF will be randomized to a flecainide (class I AAD) or sotalol (class III AAD) in order to determine if response to therapy is modified by chr4q25 SNPs using AF burden as a metric of drug efficacy. This main study, like the pilot study proposed here, will utilize a crossover design to minimize inter-individual variability and maximize statistical power to detect an interaction between chr4q25 genotype and the reduction of AF burden with flecainide vs. sotalol. After a run-in period during which the AAD will be up-titrated, subjects will be monitored with the Medtronic Reveal LINQ Insertable Cardiac Monitor (ICM) system to assess AF burden. Furthermore, subjects will be asked to complete a comprehensive, validated 20-item AF specific questionnaire (AF Effect on QualiTy-of-life [AFEQT]) at baseline, and monthly thereafter for the duration of the study. At the end of the 6-month trial period, the AAD will be discontinued and participants will be switched to the other AAD and followed for another 6-month period in a crossover trial design.

2.0 Rationale and Specific Aims

We and others have shown common SNPs at the chr4q25 locus are associated with increased risk of AF and modulate symptomatic response to AADs. Furthermore, our preliminary data suggests that there is a differential response to class I vs. class III membrane-active drugs. Here, we propose a pilot study to obtain preliminary data regarding AF burden in patients receiving AADs and to demonstrate feasibility for a future study to test the hypothesis that chr4q25 risk SNPs modulate differential response to AADs in patients with frequent symptomatic paroxysmal AF using reduction in mean AF burden as a metric of drug efficacy. Therefore, the Specific Aim of this pilot/feasibility study is to obtain preliminary data regarding AF burden in patients receiving AADs and to demonstrate feasibility for a future study to test the hypothesis that chr4q25 SNPs modulate differential response to class I vs. class III AADs in patients with frequent symptomatic AF.

3.0 Previous Human Studies

Chr4q25 SNPs modulate differential response to AADs in patients with AF In a preliminary study we addressed whether symptomatic response to AAD therapy is modulated by the 3 common AF susceptibility loci on chr4q25 (near PITX2), 16q22 (in ZFHX3), and 1q21 (in KCNN3). We studied 478 (discovery cohort) and 198 (validation cohort) age and gender matched Caucasian patients in the Vanderbilt AF Registry. Response to AAD therapy was defined as successful rhythm control if the patient remained on the same AAD therapy for a minimum of 6 months with ≥ 75% reduction in AF symptoms. Multiple clinical variables (including age, hypertension, lone AF) failed to predict response to AADs. However, a SNP at the 4q25 locus (rs10033464) was significantly associated with successful symptom control (odds ratio [OR] 2.97, 95% confidence interval [CI] 1.42-6.21, P=0.003). Furthermore, individuals who carried the 4q25 SNP responded better to class I vs. class III AADs in both the discovery and validation cohorts. These preliminary findings provide the rationale for our future studies by suggesting that common AF susceptibility variants differentially modify the response to class I vs. class III AADs in patients with frequent symptomatic AF.

4.0 Enrollment/Randomization

Patients ≥18 years of age with symptomatic paroxysmal AF will be enrolled from the Arrhythmia and Cardiology Clinics, the Adult Emergency Department, and inpatient Cardiology services at University of Illinois Medical Center. For patients with whom researchers do not have a relationship, introductions from a member of their care team will be sought prior to discussion of the study. After obtaining the permission of the patient, a member of the study team will explain the study, answer any questions, and allow sufficient time to be certain that the subject understands the study and has given their consent to participate. Consent will be documented by signing the informed consent document, a copy of which will be given to the subject.

5.0 Study Procedures

Randomization: Patients will be consented and randomized to either flecainide or sotalol for six months and then crossed-over to the alternate drug for six months, regardless of the efficacy of the first drug. Study randomization will be through http://www.randomize.net/. Each participating will have access to the randomization application and each site responsible per their local IRB regulations to maintain the randomization study list. The study will be open-label.

Baseline visit procedures: The baseline visit will take place at the AF and Cardiology Clinic at the Outpatient Care Center (OCC) of UIHHSS. This visit will involve reviewing eligibility and the consenting process. Patients will present to the OCC and be met by a study physician, who will perform a history and physical exam. A baseline 12-lead ECG will be obtained for all patients and interpreted by the study physician to verify eligibility. Patients who meet the criteria will be randomized into one of the two study medications (sotalol or flecainide), and scheduled by a study nurse to come back to UIHHSS within one week to receive the Medtronic Reveal ICM implantation and administered the initial dose of study drug.

For patients randomized to start sotalol first, they will be scheduled by the study nurse to return to UIH in approximately 1 week to be admitted for up to 72 hours, which is routinely done for sotalol administration. The designated cardiology/AF nurse will schedule this admission after the consenting/baseline visit is completed in the clinic. At the second visit, once inclusion and exclusion criteria are confirmed again for continued eligibility, a peripheral intravenous catheter will be placed, and blood will be drawn for a basic metabolic panel (BMP), particularly potassium (K+) and creatinine (Cr). This is routinely done for patients hospitalized for initiation of sotalol. The study physician will determine the initial sotalol dose (80 - 120mg twice a day by mouth) based on Cr CL.

Two hours after the first dose of study drug is given a 12-lead ECG will be recorded and interpreted by the study physician. If the QTc is >500 msec, the sotalol dose will be reduced under the direction of the study physician. Patients will be admitted for continuous telemetric monitoring and will remain in UIH until the 5th dose is administered as long as the physician confirms eligibility with each dose. Additional 12-lead ECGs will be obtained two hours after the 3rd and 5th doses of sotalol to assess QTc duration. The BMP will also be drawn to routinely monitor the subject's K+ and Cr. If the QTc duration remains >500 msec even after adjustment of the sotalol dose, the drug will be stopped and the patient will be excluded from the study. If the QTc remains ≤500 msec after the 5th dose of sotalol, the patient will be discharged to home.

Intravenous sotalol rapid initiation will be also available to study participants. Patients admitted to University of Illinois Hospital and Clinics (Hospital) to initiate treatment are admitted to the cardiology service and located on 6 West Step-Down or 7 East Step-Down nursing unit with continuous cardiac telemetry monitoring. See study addendum for intravenous sotalol rapid initiation clinical care guideline.

A phone call will be made by the study coordinator or study physician 3 days after discharge to check subject's status and ensure they are tolerating sotalol and are not experiencing any untoward side effects.

Patients randomized to flecainide at the baseline visit will initially be scheduled for follow up at the UIH Electrophysiology Laboratory within one week. At the second visit, once inclusion and exclusion criteria are confirmed again for continued eligibility, a LINQ ICM will be inserted. The patient will be observed for two hours after the ICM insertion. During this time, an ECG will be performed and a quality of life (QoL) questionnaire will be administered. After 2 hours of observation after ICM insertion, the 1st dose of flecainide will be administered (50-100mg at physician's discretion). As per guidelines for flecainide, subjects will also concomitantly be started on either beta blockers (25 mg by mouth once a day) or diltiazem (120 mg long-acting by mouth once a day) based on the patient's tolerability. An AV nodal blocker like beta blockers and diltiazem is often co-prescribed with flecainide to prevent the development of 1:1 conducted atrial flutter.

After the 1st dose of flecainide (+beta blockers /diltiazem), there will be 2 hours of observation to capture any outcomes/adverse reactions, and another ECG will be done to examine the PR interval and QRS duration. The study physician will review these and decide if patient is eligible to continue and make any adjustments as needed. A 3-day phone call will be made by the study physician or another member of the research team to check subject's status and obtain any outcomes.

End of study procedures: Patients will be scheduled for a clinic visit with their primary cardiac arrhythmia physician to coincide with the termination of the study (12 months). A study physician will also be available to conduct a brief patient interview, pill count, and ICM interrogation. All pertinent clinical data including AF burden on each AAD, maximal tolerated dose, and any reported side effects will be given to the primary arrhythmia physician to aide in clinical decision making about future AAD

Early study termination, early crossover, and procedures to treat persistent AF: Based on our prior clinical experience, a proportion of patients (20 to 30%) are expected to experience residual symptomatic episodes of AF while taking either or both study AADs. Usually these episodes will be less bothersome or lengthy. Patients will be encouraged to continue the study protocol if possible. However, a smaller proportion of patients might have intolerable symptoms necessitating an unscheduled change in therapy. The study team will work with the primary cardiac electrophysiologist to facilitate any necessary change in therapy. An early crossover to the alternative study AAD will be encouraged over a change to a non-study AAD when possible. A change in therapy to a non-study AAD or AF ablation procedure will be allowed when necessary. In addition, if patients acquire persistent AF during the course of the study, electrical cardioversion will be allowed and will be coordinated by the study team and the primary cardiac electrophysiologist. AF burden data for patients deviating from the study protocol will be analyzed using an "on treatment" analysis. In other words, the AF burden will be calculated per day that patients are on each study AAD. Patients will also be allowed to withdraw from the study for personal or other reasons at any time. Patients are volunteering their time, so they reserve the right to withdraw from the study at any point.

Insertable cardiac monitor management after study termination: At the conclusion of the twelve-month study, patients will be given the option to remove or retain the ICM. We anticipate that most patients and their primary arrhythmia physicians will opt to retain the device to allow for continued cardiac monitoring, which is not only useful to gauge response to AAD therapy but also frequently used to monitor AF recurrence for patients undergoing catheter ablation. If the ICM is retained, its management, including removal, will be transferred to the primary electrophysiologist. Patients wishing to have the ICM removed at the end of the study period will be scheduled for an outpatient visit to the UIH EP Laboratory for removal by a study physician.

Primary end point and its determination: The primary endpoint will be mean AF burden over six months as measured by the Medtronic Reveal LINQ ICM system. All patients are scheduled to remain in the study for 12 months. The FDA-approved Medtronic Reveal LINQ ICM system is able to continuously monitor the heart through a single-lead ECG and has a specific algorithm that detects AF by evaluating the irregularity of R-R intervals.The device is able to correctly classify AF in 96.1% of patients and correctly exclude AF in 97.4% of subjects.The device is able to monitor the heart for up to 3 years and is compatible with the Medtronic CareLink Network remote monitoring system. This system allows the treating physician to download device and diagnostic data through a secure network. Patients transmit data manually after the device indicates that one of the alert criteria have been met. The occurrence of symptoms with the AF episode will be recorded, but both asymptomatic and symptomatic AF will be included in the primary endpoint measurement of AF burden.

For the primary analysis, AF burden will begin to be tabulated after an initial run in period for each study drug. For patients starting sotalol, the run-in period will coincide with the first 5 doses (60 hours). For patients starting flecainide, the run-in period will last until a dose of at least 200 mg per day (in divided doses) is achieved, unless a smaller dose is the maximally tolerated dose. Ideally, this will be achieved within 3-4 days after initiation of flecainide. If, during the course of the study, a patient develops persistent AF, a cardioversion will be scheduled in coordination with the patient's primary electrophysiologist. The patient will then be switched to the other study drug. In case of such an occurrence, AF burden will be tabulated using an "on treatment" analysis. Conditions for which a patient will be withdrawn from the study and data censored will be discontinuation of AAD therapy, initiation of amiodarone, AF ablation or AV node ablation/permanent pacing, loss to follow-up, elective withdrawal from the study, or death.

Blood processing, DNA extraction, and genotyping: Blood samples will be drawn into ethylenediamenetetraacetic acid (EDTA) tubes and immediately refrigerated at 4° C. Plasma will be separated by centrifugation and stored at -80° C. DNA will be extracted from the buffy coat using a commercially available kit (Qiagen Puregene, Valencia, California) and stored at -20° C. Study participants will be genotyped for three common chr4q25 SNPs (rs2200733, rs17570669, and rs3853445) using Sanger sequencing.

6.0 Risks

Risks will be minimized by performing study procedures in the UIHHSS EP Laboratory. A complete history and physical examination will be performed to ensure that subjects fulfill the entry criteria as defined. All identifying documents and data collected as a result of this study will be retained by the investigator. Data will be entered into the secure Research Electronic Data Capture (REDCap) database. Access to this material will be available only to the research investigator and his staff. If results of this study are to be published, only randomized code numbers will be used for identification purposes. Participants will not be identified by name.

Risks associated with the Medtronic Reveal LINQ ICM: Risks associated with insertion of the ICM include pain and discomfort, bleeding, bruising, hematoma, infection, and an allergic reaction to the skin prep or lidocaine used for local anesthesia. There is a very small risk of long-term discomfort associated with having the device. According to the manufacturer, the ICM is fully MRI-compatible immediately after implantation.

Risks associated with sotalol: Therapeutic doses of sotalol range from 160 mg to 240 mg per day. Common side effects of sotalol therapy include bradycardia (13% to 16%), chest pain (3% to 16%), palpitations (14%), fatigue (20%), dizziness (20%), lightheadedness (12%), weakness (13%), dyspnea (21%), edema (8%), hypotension (6%), proarrhythmia (5%), syncope (5%), heart failure (5%), torsade de pointes (dose related; 1% to 4%), peripheral vascular disorders (3%), ventricular tachycardia worsened (1%), QTc interval prolongation (dose related), headache (8%), sleep problems (8%), mental confusion (6%), anxiety (4%), depression (4%), rash (5%), sexual side effects (3%), nausea/vomiting (10%), diarrhea (7%), stomach discomfort (3% to 6%), flatulence (2%), impotence (2%), bleeding (2%), extremity pain (7%), paresthesia (4%), back pain (3%), visual problems (5%), upper respiratory problems (5% to 8%), and asthma (2%). Rare (<1%) side effects of therapeutic doses of sotalol include alopecia, bronchiolitis obliterans with organized pneumonia (BOOP), cold extremities, diaphoresis, eosinophilia, leukocytoclastic vasculitis, leukopenia, paralysis, phlebitis, photosensitivity reaction, pruritus, pulmonary edema, Raynaud's phenomenon, red crusted skin, retroperitoneal fibrosis, elevated liver transaminases, thrombocytopenia, and vertigo.

Risks associated with flecainide: Therapeutic doses of flecainide range from 200 mg to 300 mg per day. Common side effects of flecainide therapy include dizziness (19% to 30%), visual disturbances (16%), dyspnea (10%), palpitations (6%), chest pain (5%), edema (3.5%), tachycardia (1% to 3%), proarrhythmia (4% to 12%), sinus node dysfunction (1.2%), syncope, headache (4% to 10%), fatigue (8%), nervousness (5%), fever, malaise, hypoesthesia, paresis, ataxia, vertigo, somnolence, tinnitus, anxiety, insomnia, depression, rash (1% to 3%), nausea (9%), constipation (1%), abdominal pain (3%), anorexia (1% to 3%), diarrhea (0.7% to 3%), tremor (5%), weakness (5%), paresthesia (1%), diplopia (1% to 3%), and blurred vision. Rare (< 1%) side effects include alopecia, altered pacing threshold, amnesia, angina, AV block, bradycardia, bronchospasm, heart failure, corneal deposits, depersonalization, euphoria, exfoliative dermatitis, granulocytopenia, heart block, increased PR interval, leukopenia, metallic taste, neuropathy, paradoxical increase in ventricular rate in atrial fibrillation/flutter, paresthesia, photophobia, pneumonitis, pruritus, increased QRS duration, swollen lips/tongue/mouth, tardive dyskinesia, thrombocytopenia, urinary retention, urticaria, and ventricular arrhythmias.

Risks associated with oral beta blockers use: Therapeutic dose of beta blockers ranges from 50 mg to 200 mg per day. Common side effects of chronic beta blockers therapy include tiredness (26%), dizziness (13%), depression (12%), cold, tingling, or numbness in the hands or feet (12%), and shortness of breath (6%). Other common adverse effects of beta blockers include slow heart rate (bradycardia), a decrease in blood pressure when going from a lying-down or sitting position to standing, a spinning sensation (vertigo), lightheadedness, diarrhea, and nausea. We will use a low dose of beta blockers (25 mg) in this study to minimize the risk of occurrence of these adverse effects. Rare (< 1%) side effects of therapeutic doses of beta blockers include an increase in liver enzymes, allergic reactions, headache, impotence (also known as erectile dysfunction), Peyronie's disease, worsening of psoriasis, reversible hair loss, vision problems, dry mouth, Raynaud's phenomenon, unexplained rash, and dry eyes. These adverse effects are not anticipated with a single low dose of beta blockers that will be administered to our volunteers. Beta blockers can rarely cause an allergic reaction (<1%) that manifests as rash, itching, swelling, severe dizziness, or trouble breathing. Any subject with a previous history of allergy or intolerance to beta-blockers will be excluded from the study.

Risks associated with oral diltiazem use: The therapeutic dose of diltiazem ranges from 120 mg to 480 mg per day. Common side effects of chronic diltiazem therapy include edema (2% to 15%), headache (5% to 12%), AV block (first degree 2% to 8%), bradycardia (2% to 6%), hypotension (2% to 4%), vasodilation (2% to 3%), extrasystoles (2%), flushing (1% to 2%), palpitation (1% to 2%), dizziness (3% to 10%), nervousness (2%), rash (1% to 4%), gout (1% to 2%), dyspepsia (1% to 6%), constipation (<2% to 4%), vomiting (2%), diarrhea (1% to 2%), weakness (1% to 4%), myalgia (2%), rhinitis (<2% to 10%), pharyngitis (2% to 6%), dyspnea (1% to 6%), bronchitis (1% to 4%), cough (≤3), and sinus congestion (1% to 2%). Rare (< 1%) side effects of diltiazem include an increase in alkaline phosphatase, allergic reaction, increase in liver transaminases, amblyopia, amnesia, arrhythmia, AV block (second or third degree), bundle branch block, heart failure, depression, dysgeusia, extrapyramidal symptoms, gingival hyperplasia, hemolytic anemia, petechiae, photosensitivity, Stevens-Johnson syndrome, syncope, tachycardia, thrombocytopenia, tremor, and toxic epidermal necrolysis.

Risks associated with venipuncture: Potential problems related to establishing an intravenous access include pain, bleeding, hematoma, fainting, and rarely infection at the venipuncture site.

7.0 Reporting of Adverse Events or Unanticipated Problems Involving Risk to Participants or Others

All adverse events will be reported to the institutional review board (IRB) within five business days as required by institutional policy. A serious adverse event is defined as an untoward medical occurrence that results in death, is life-threatening, requires hospitalization, results in persistent or significant disability, or requires intervention to prevent permanent disability or death. Other untoward medical occurrences that do not meet the above criteria will be classified as adverse events. Study personnel who are administering the research protocol in the UIH EP Laboratory will monitor for adverse events, with the assistance of the designated nursing staff. All suspected or confirmed adverse events will promptly be reported to the PI, who will collect data on these occurrences. The PI will report serious adverse events to the IRB within 5 days of being notified.

8.0 Study Withdrawal/Discontinuation

Participation in the study is strictly voluntary, and patients will be able to withdraw at any time. Following the subject's withdrawal, any samples collected will be destroyed and not analyzed further, although any analyzed data will be maintained.

9.0 Statistical Considerations

Sample size: The primary outcome will be comparison of mean reduction in AF burden when treated with flecainide vs. sotalol for 6 months each. Based on our pilot study, the mean AF burden on flecainide was 20±14% (SD). As the minor allele frequency (MAF) of rs10033464 is ~12%, the ratio of carriers to non-carriers is ~1:8. A mean reduction in AF burden of 10% in chr4q25 AF risk allele vs. WT allele carriers may be clinically meaningful assuming that half of the patients will receive flecainide first and the other half sotalol first. In order to detect at least a 50% difference in AF burden on the two AADs (absolute difference of 10%), the study requires a total of 162 patients to achieve 80% power in detecting the difference. Sample size computation was performed using an approximate t-test with pooled variance estimate that compared mean reduction in AF burden over 6 months with a 2-sided 5% significance level. SD of the mean reduction in AF burden was estimated to be 14% (based on the pilot study) assuming a correlation of 10% among repeated measures and a 20% drop-out rate.

Statistical analysis: The primary study endpoint will be AF burden (the proportion of time a patient is in AF) and will be calculated for each subject while being treated with flecainide and sotalol. For the primary analysis, we will test the hypothesis that the chr4q25 AF risk allele (rs10033464) modulates the treatment effect difference between flecainide and sotalol. The average burden difference on the two treatments between patients carrying the AF risk allele and those carrying the WT allele will be calculated and the hypothesis will be tested using an approximate t-test based on the standardized score (divided by its standard error). No adjustment of covariates such as age and gender will be required because the cross-over design controls for such variables. The analysis will be performed both on the patients who complete the study and on all patients intended to treat with outcomes of the drop-outs imputed. Conventional imputations using last-observation-carry-forward, as well as model-based imputations will be performed to assess the robustness of the findings based on patients who complete the study.

A secondary analysis using a mixed effects model will be performed treating the AF burden score measurement over the treatment course of a patient as longitudinal data. Clinical covariates that may affect AF burden (age, male sex, diabetes mellitus, HTN, valvular disease, coronary artery disease, heart failure, and obesity) will be included in the mixed effects model to examine the effects of a patient's profile, AAD therapy, as well as their interactions with the AF burden scores. [In addition, a number of exploratory analyses will be performed on other AF risk alleles, particularly the other 3 most common chr4q25 AF SNPs (rs2200733, rs17570669, rs3853445) associated with AF in EAs26 to determine if any of them modulate response to flecainide and sotalol, using the same test for the primary analysis based on the AF burden scores. Specifically, the analysis will explore (a) the joint effect of all 4 AF SNPs using a multivariate test; (b) the effects of individual SNPs if the global test detects statistical significance; and (c) the effect of collapsed genetic scores created by coding each patient's genotype as the sum number of variant alleles carried across all 4 AF SNPs. We expect that the chr4q25 SNPs may demonstrate a sufficiently strong association with AF burden to drive the effect observed in our combined analysis of all 4 SNPs. As is common practice in genetic analysis of complex diseases like AF, all analyses will be tested using both dominant and additive genetic models.

10.0 Privacy/Confidentiality Issues

All research hard copy records will be stored in a locked cabinet within a locked office with access only to the research personnel. Digitalized ECG recordings will be de-identified and stored in a password-protected electronic database. Only the investigators and members of the study team will have access to the code key.

A possible risk of the research is that information about a patient's health might become known to individuals outside the research. The investigators have put in place measures to minimize this risk as described below.

All identifying documents, data, and specimens collected as a result of this study will be retained by Dr. Darbar. Data will be entered by hand onto a blank copy of the data collection packet, which was generated on the secure Research Electronic Data Capture (REDCap) database. The more comprehensive study in the future will most likely use the REDCap database directly online for convenience. Access to this material will be available only to the research investigator and his staff. If results of this study are to be published, only randomized code numbers will be used for identification purposes.

Completing the QoL questionnaires will not pose greater loss of confidentiality as all forms will be kept with the subject file. These files will be safely stored in Dr. Darbar's research offices, in a filing cabinet that is locked. Only the research staff and Dr. Darbar have access to this locked cabinet. The information will only remain with the designated research staff. If results of this study are to be published, only randomized code numbers of subjects will be used to protect their identity. Participants will not be identified by name or any study identifiers.

11.0 Follow-up and Record Retention

We expect that the study will span a period of 12 months. All data will be archived and stored indefinitely.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* History of typical or early-onset symptomatic (≥2 episodes/month) paroxysmal/persistent AF
* ECG that was recorded within 1 month of randomization showing AF
* Eligible for both Flecainide(Class I) and Sotalol (Class III) AAD
* Able to give informed consent

Exclusion Criteria:

* Permanent AF or isolated atrial flutter
* Cardiac or thoracic surgery within the previous 6 months
* Previous use of amiodarone other than short-term use (e.g. for an acute arrhythmia in hospital)
* Medical condition that is likely to be fatal in less than one year
* A history of prior AF ablation
* Have already been tried on 2 or more AADs in the past for AF
* Creatinine clearance <40 ml/min
* Left ventricular ejection fraction < 50%
* Contra-indication to a Class I AAD e.g., structural heart disease, or history of MI
* Contra-indication to a Class III AAD, e.g., congenital or acquired long QT syndrome with QTc>480 ms in females and >460 ms in males at baseline
* A reversible cause of AF (e.g., hyperthyroidism)
* Females who are pregnant or nursing
* History of severe AV node dysfunction unless an electronic pacemaker is present
* First- or second-degree relative has already participated in the study
* Unable to adhere to study procedures that are strictly for research purposes

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2020-12-31 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
AF burden (Percent of time subject is in atrial fibrillation) | 12 months
  Subjects will be monitored with the Medtronic Reveal LINQ Insertable Cardiac Monitor (ICM) system to assess AF burden. The device will be programmed to optimize the memory for storing AF episode.

SECONDARY OUTCOMES:
AF Effect on QualiTy-of-life [AFEQT] | 12 months
  Quality of life assessment: Patients will be asked to fill out the AFEQT quality of life questionnaire baseline (study randomization), two, four, six, eight, ten, and 12 months (completion of the study). The questionnaire at the end of the 6rd month will be administered just prior to stopping the first study drug. The validated questionnaire is comprised of 20 questions about AF symptoms with answers given on a Likert scale. The questionnaire will be provided to the patients in paper format either in person or by mail, as applicable. A follow-up phone call will be made to each patient to ensure that the questionnaire is completed and returned.
  The responses on the 20-item AFEQT are scored on a 1 to 7 Likert scale ranging from 1: "Not at all", 2:" Hardly", 3: "A little ", 4: "Moderately", 5: "Quite a bit, 6:" Very" to 7: "Extremely".
  A total score of 0 corresponds to complete disability, while a score of 100 describes the highest level of QualiTy-of-life

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Jesse Brown VA Medical Center, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois